CLINICAL TRIAL: NCT00285376
Title: A Randomized, Double-Blind, Placebo Controlled Study Assessing the Efficacy and Safety of Vilazodone and Discovering Genetic Markers Associated With Response in Patients With Major Depressive Disorder
Brief Title: Effectiveness Study of Vilazodone to Treat Depression and to Discover Genetic Markers Associated With Response
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genaissance Pharmaceuticals (Industry)
Responsible Party: Carol Reed, MD, Genaissance Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNSC-04-DP-02
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Depressive Disorder, Major
Keywords: Depression. Genetics, Pharmacogenetics
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vilazodone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): vilazodone
  Interventions: Drug: vilazodone
- 2 (Placebo Comparator)
  Interventions: Drug: vilazodone

INTERVENTIONS:
Drug: vilazodone — titration to 40mg tablets qd for 8 weeks
  Other Names: EMD 68843, SB-659746

SUMMARY:
This study is designed to determine the safety and effectiveness of vilazodone for major depressive disorder and to discover genetic markers associated with response. This study will enroll approximately 400 patients.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, multicenter, 8-week, clinical trial is designed to assess the efficacy and safety of vilazodone and to discover genetic markers of treatment response associated with vilazodone use in adult patients diagnosed with MDD by the DSM-IV-TR criteria. This study will enroll approximately 400 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18-65 years of age, inclusive.
* A diagnosis of MDD, single episode or recurrent, according to DSM-IV-TR (296.2/296.3) with a current Major Depressive Episode of less than two year's duration with a minimum duration of at least 4 weeks.
* HAM-D score ≥ 22.
* HAM-D item 1 (depressed mood) score ≥ 2.
* Patients must be able to provide written informed consent to participate before beginning any trial related activities.
* Patients must be able to speak, read and understand English and possess the ability to respond to questions and follow simple instructions.

Exclusion Criteria:

* A current (or within 6 months prior to the Screening Visit) Axis I disorder of Post Traumatic Stress Disorder, Eating Disorder, Obsessive Compulsive Disorder (Generalized Anxiety Disorder, Social Phobia or Simple Phobia will be allowed).
* A history of schizophrenia, schizoaffective disorder or bipolar I or II disorder (with a history of hypomanic or manic episodes).
* DSM-IV-TR criteria for substance abuse (alcohol or drugs) within 3 months prior to Screening Visit or substance dependence within 6 months prior to the Screening Visit.
* Criteria for any of the following DSM-IV-TR MDD Specifiers: [a] With Catatonic Features; [b] With Postpartum Onset; [c] With Seasonal Pattern.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2006-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
MADRS | 8 weeks

SECONDARY OUTCOMES:
HAM-D | 8 weeks
CGI | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carol Reed, M.D., Study Director — Genaissance Pharmaceuticals
Locations (15):
- United States (15):
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - Pharmacology Research Institute, Northridge, California
  - Pharmacology Research Institute, Riverside, California
  - Atlanta Institute of Medicine & Research, Atlanta, Georgia
  - Atlanta Institute of Medicine & Research, Marietta, Georgia
  - Summit Research Network (Michigan), Inc., Farmington Hills, Michigan
  - Summit Research Network (Michigan), Inc., Flint, Michigan
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - University of Pennsylvania Department of Psychiatry Mood and Anxiety Disorders Section, Philadelphia, Pennsylvania
  - Southeast Health Consultants, LLC, Charleston, South Carolina
  - University of Utah health Services Center Dept. of Psychiatry Mood and Anxiety Disorders, Salt Lake City, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network (Seattle) LLC, Seattle, Washington

REFERENCES:
- [Derived] Kornstein S, Chang CT, Gommoll CP, Edwards J. Vilazodone efficacy in subgroups of patients with major depressive disorder: a post-hoc analysis of four randomized, double-blind, placebo-controlled trials. Int Clin Psychopharmacol. 2018 Jul;33(4):217-223. doi: 10.1097/YIC.0000000000000217. PMID 29608461
- [Derived] Culpepper L, Mathews M, Ghori R, Edwards J. Clinical relevance of vilazodone treatment in patients with major depressive disorder: categorical improvement in symptoms. Prim Care Companion CNS Disord. 2014;16(1):PCC.13m01571. doi: 10.4088/PCC.13m01571. Epub 2014 Jan 30. PMID 24940525
- [Derived] Jain R, Chen D, Edwards J, Mathews M. Early and sustained improvement with vilazodone in adult patients with major depressive disorder: post hoc analyses of two phase III trials. Curr Med Res Opin. 2014 Feb;30(2):263-70. doi: 10.1185/03007995.2013.855188. Epub 2013 Oct 31. PMID 24127687
- [Derived] Clayton AH, Kennedy SH, Edwards JB, Gallipoli S, Reed CR. The effect of vilazodone on sexual function during the treatment of major depressive disorder. J Sex Med. 2013 Oct;10(10):2465-76. doi: 10.1111/jsm.12004. Epub 2012 Dec 6. PMID 23216998
- [Derived] Reed CR, Kajdasz DK, Whalen H, Athanasiou MC, Gallipoli S, Thase ME. The efficacy profile of vilazodone, a novel antidepressant for the treatment of major depressive disorder. Curr Med Res Opin. 2012 Jan;28(1):27-39. doi: 10.1185/03007995.2011.628303. Epub 2011 Nov 23. PMID 22106941
- [Derived] Rickels K, Athanasiou M, Robinson DS, Gibertini M, Whalen H, Reed CR. Evidence for efficacy and tolerability of vilazodone in the treatment of major depressive disorder: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2009 Mar;70(3):326-33. doi: 10.4088/jcp.08m04637. Epub 2009 Mar 10. PMID 19284933